CLINICAL TRIAL: NCT01666067
Title: Vascular and Metabolic Effects of Vytorin vs Simvastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Kwang Kon Koh, professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMC-201110
Record Dates: First submitted 2012-08-15; First posted 2012-08-16 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2012-08

CONDITIONS: Hypercholesterolemia
Keywords: insulin resistance
MeSH Terms: conditions — Hypercholesterolemia; Insulin Resistance | interventions — Ezetimibe, Simvastatin Drug Combination; Simvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Active Comparator): placebo
  Interventions: Drug: placebo
- vytorin (Active Comparator): vytorin
  Interventions: Drug: vytorin
- simvastatin (Active Comparator): simvastatin
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: placebo
  Arms: placebo
Drug: vytorin
  Arms: vytorin
Drug: simvastatin
  Arms: simvastatin

SUMMARY:
The investigators hypothesize that vytorin will improve insulin resistance compared with simvastatin

ELIGIBILITY:
Inclusion Criteria:

* hypercholesterolemic patients (LDL cholesterol levels>100 mg/dl)

Exclusion Criteria:

* overt liver disease, chronic renal failure, hypothyroidism, myopathy, uncontrolled diabetes (HbA1c > 9%), severe hypertension, stroke, acute coronary events, coronary revascularization within the preceding 3 months, or alcohol abuse

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
flow-mediated dilation | 8 weeks of treatment

SECONDARY OUTCOMES:
insulin resistance | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea